CLINICAL TRIAL: NCT06267872
Title: A Phase 1 Clinical Trial in Adult Participants Without HIV and in Overall Good Health to Evaluate the Safety and Immunogenicity of CD4BS CH505M5 Pr-NP1 Followed by CH505 TF chTrimer Boost Both Adjuvanted With Either Lipid Nanoparticles (LNPs) or 3M-052-AF + Alum
Brief Title: A Clinical Trial in Adult Participants Without HIV and in Overall Good Health to Evaluate the Safety and Immunogenicity of CD4BS CH505M5 Pr-NP1 Followed by CH505 TF chTrimer Boost Both Adjuvanted With Either Lipid Nanoparticles (LNPs) or 3M-052-AF + Alum
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA Clinical Hold
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency); Duke University (Other); Access to Advanced Health Institute (AAHI) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 309
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: HIV
MeSH Terms: interventions — Product Labeling; aluminum sulfate; Aluminum Hydroxide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A - Group 1 (Experimental): • 60 mcg of CD4BS CH505M5 Pr-NP1, to be administered as two 0.5 mL doses intramuscularly at months 0, 2, and 4.
  Interventions: Biological: CD4BS CH505M5 Pr-NP1
- Part B - Group 2 (Experimental): * 60 mcg of CD4BS CH505M5 Pr-NP1, admixed with 1.0 mg of ACU-026-001-1 adjuvant to be administered as two 0.5 mL doses intramuscularly at months 0, 2, and 4
  * Followed by 300 mcg of CH505TF chTrimer, admixed with 1.0 mcg of ACU-026-001-1 adjuvant to be administered at months 6 and 8.
  Interventions: Biological: CD4BS CH505M5 Pr-NP1; Biological: CH505TF chTrimer; Biological: ACU-026-001-1 (labeled as empty LNP)
- Part B - Group 3 (Experimental): * 60 mcg of CD4BS CH505M5 Pr-NP1, admixed with 2.0 mg of ACU-026-001-1 adjuvant to be administered as two 0.5 mL doses intramuscularly at months 0, 2, and 4
  * Followed by 300 mcg of CH505TF chTrimer, admixed with 2.0 mg of ACU-026-001-1 adjuvant to be administered at months 6 and 8.
  Interventions: Biological: CD4BS CH505M5 Pr-NP1; Biological: CH505TF chTrimer; Biological: ACU-026-001-1 (labeled as empty LNP)
- Part B - Group 4 (Experimental): * 60 mcg of CD4BS CH505M5 Pr-NP1, admixed with 5 mcg of 3M-052-AF adjuvant along with 500 mcg of Alum to be administered as two 0.5 mL doses intramuscularly at months 0, 2, and 4
  * Followed by 300 mcg of CH505TF chTrimer, admixed with 5 mcg of 3M-052-AF adjuvant along with 500 mcg of Alum to be administered to be administered at months 6 and 8.
  Interventions: Biological: CD4BS CH505M5 Pr-NP1; Biological: CH505TF chTrimer; Biological: 3M-052-AF (labeled as AP 60-702); Biological: Aluminum Hydroxide Suspension (Alum)
- Part C - Group 5 (Experimental): Low dose:
  * 100 mcg of CD4BS CH505M5 Pr-NP1, admixed with 1.0 mg of ACU-026-001-1 adjuvant to be administered as two 0.5 mL doses intramuscularly at months 0, 2, and 4,
  * Followed by 300 mcg of CH505TF chTrimer, admixed with 1mg empty LNP adjuvant to be administered at months 6 and 8.
  OR,
  High Dose:
  * 100 mcg of CD4BS CH505M5 Pr-NP1, admixed with 2.0 mg of ACU-026-001-01 adjuvant to be administered as two 0.5 mL doses intramuscularly at month 0, 2, and 4,
  * Followed by 300 mcg of CH505TF chTrimer, admixed with 2.0 mg of ACU-026-001-1 adjuvant to be administered at months 6 and 8.
  Interventions: Biological: CD4BS CH505M5 Pr-NP1; Biological: CH505TF chTrimer; Biological: ACU-026-001-1 (labeled as empty LNP)
- Part C - Group 6 (Experimental): * 100 mcg of CD4BS CH505M5 Pr-NP1, admixed with 3 mcg of 3M-052-AF adjuvant along with 500 mcg of Alum to be administered as two 0.5 mL doses intramuscularly at months 0, 2, and 4,
  * Followed by 300 mcg of CH505TF chTrimer, admixed with 3 mcg of 3M-052-AF adjuvant along with 500 mcg of Alum to be administered to be administered at months 6 and 8.
  Interventions: Biological: CD4BS CH505M5 Pr-NP1; Biological: CH505TF chTrimer; Biological: 3M-052-AF (labeled as AP 60-702); Biological: Aluminum Hydroxide Suspension (Alum)
- Part C - Group 7 (Experimental): * 100 mcg of CD4BS CH505M5 Pr-NP1, admixed with 5 mcg of 3M-052-AF adjuvant along with 500 mcg of Alum to be administered as two 0.5 mL doses intramuscularly at months 0, 2, and 4
  * Followed by 300 mcg of CH505TF chTrimer, admixed with 5 mcg of 3M-052-AF adjuvant along with 500 mcg of Alum to be administered to be administered at months 6 and 8.
  Interventions: Biological: CD4BS CH505M5 Pr-NP1; Biological: CH505TF chTrimer; Biological: 3M-052-AF (labeled as AP 60-702); Biological: Aluminum Hydroxide Suspension (Alum)

INTERVENTIONS:
Biological: CD4BS CH505M5 Pr-NP1 — A ferritin NP expressing 8 copies of an HIV-1 Env protein trimer. To be administered intramuscularly (IM).
Biological: CH505TF chTrimer — A stabilized chimeric SOSIP Env trimer protein with the N-terminal sequence of CH505 TF gp120 Env transplanted into the BG505 SOSIP sequence. To be administered IM.
  Arms: Part B - Group 2; Part B - Group 3; Part B - Group 4; Part C - Group 5; Part C - Group 6; Part C - Group 7
Biological: 3M-052-AF (labeled as AP 60-702) — An aqueous formulation (AF) of the small molecule imidazoquinoline immune response modifier (IRM) 3M-052; toll-like receptor (TLR)7/8 agonist.
  Arms: Part B - Group 4; Part C - Group 6; Part C - Group 7
Biological: Aluminum Hydroxide Suspension (Alum) — Alum to be administered IM as 500 mcg (aluminum content) admixed with 3M-052-AF (5 mcg) along with CD4BS CH505M5 Pr-NP1 and CH505 TF chTrimer.
  Other Names: Alhydrogel
  Arms: Part B - Group 4; Part C - Group 6; Part C - Group 7
Biological: ACU-026-001-1 (labeled as empty LNP) — An AF consisting of 4 lipid components.
  Arms: Part B - Group 2; Part B - Group 3; Part C - Group 5

SUMMARY:
This is a multicenter, open-label, phase 1 clinical trial to test two human immunodeficiency virus (HIV) vaccines with two adjuvants. An adjuvant is an ingredient used with some vaccines that may help people make an immune response. HIV is the virus that causes acquired immunodeficiency syndrome (AIDS).

About 42 people will take part in the HVTN 309 clinical trial. This clinical trial will take place at multiple sites in the US and South Africa and the clinical trial is divided into 3 parts: Part A, Part B and Part C. About 3 people will participate in Part A of this study. After results from Part A are reviewed, it will be determined whether or not Part B and Part C of the clinical trial will proceed.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to complete the informed consent process, including an Assessment of Understanding (AoU): Volunteer demonstrates an understanding of this study and completes a questionnaire prior to signing the informed consent form(s) with verbal demonstration of understanding of questionnaire items that were answered incorrectly.
2. 18 to 55 years old, inclusive, on day of enrollment.
3. Available for clinic follow-up through the last clinic visit, willing to undergo FNA and leukapheresis (for Part C only), and willing to be contacted 12 months after the last study-product administration.
4. Agrees not to enroll in another study of an investigational agent during participation in the trial. If a potential participant is already enrolled in another clinical trial, approvals from the other trial sponsor and the HVTN 309 PSRT are required prior to enrollment into HVTN 309.
5. In good general health according to the clinical judgment of the site investigator.
6. Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator.
7. Assessed by clinical staff as having a low likelihood of acquiring HIV per guidelines and agrees to discuss their potential for HIV acquisition, agrees to risk-reduction counseling, and agrees to avoid behaviors associated with a higher likelihood of acquiring HIV through the final study visit. Low likelihood may include persons stably taking pre-exposure prophylaxis (PrEP).
8. Hemoglobin (Hgb):

   * ≥ 11.0 g/dL for AFAB volunteers
   * ≥ 13.0 g/dL for cisgender AMAB volunteers and for transgender men who have been on hormone therapy for more than 6 consecutive months
   * ≥ 12.0 g/dL for transgender women who have been on hormone therapy for more than 6 consecutive months
   * For transgender volunteers who have been on hormone therapy for less than 6 consecutive months, determine Hgb eligibility based on their sex assigned at birth.
9. WBC count = 2,500 to 12,000/mm3 (WBC over 12,000/mm3 is not exclusionary if further evaluation shows general good health and if PSRT approval is granted).
10. Platelets = 125,000 to 550,000/mm3.
11. ALT < 2.5 x upper limit of normal (ULN) based on the institutional normal range.
12. Serum creatinine ≤ 1.1 x ULN based on the institutional normal range.
13. For Part C, total serum calcium level of > 8.5 mg/dL.
14. Systolic blood pressure of 90 to <140 mmHg and diastolic blood pressure of 50 to <90 mmHg at screening visit. The average blood pressure between the screening visit and the enrollment visit must be below 140 mmHg systolic and 90 mmHg diastolic. A single measurement greater than or equal to 160 systolic mmHg or 100 mmHg diastolic during the current study evaluation is exclusionary.
15. Negative HIV test results by one of the following options:

    For US volunteers:
    * US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA)
    * Chemiluminescent microparticle immunoassay (CMIA)
    * Two negative results on HIV rapid tests (one of which must be FDA-approved CMIA)

    For non-US volunteers:
    * A negative European Conformity (CE)-marked EIA
    * A CMIA
    * A negative result on two HIV rapid tests (one of these rapid tests must be CE-marked)
16. Negative for anti-Hepatitis C virus (HCV) Abs (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV Abs are detected.
17. Negative for Hepatitis B surface Ag.
18. For AFAB volunteers or volunteers who were intersex at birth and are capable of becoming pregnant (hereafter referred to as "persons of pregnancy potential"):

    * Must agree to use effective means of contraception from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.
    * Must have a negative beta human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on day of enrollment.
19. AFAB volunteers or volunteers who were intersex at birth must agree to not seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.

Exclusion Criteria:

1. Volunteer who is breastfeeding or pregnant.
2. Body mass index (BMI) ≥ 40. Enrollment of individuals with BMI ≥ 40, whom the site investigator assesses are in good health, may be considered by PSRT approval.
3. Diabetes mellitus (DM). Type 2 DM controlled with diet alone (and confirmed by HgbA1c ≤ 8% within the last 6 months) or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with Type 2 DM that is well controlled on hypoglycemic agent(s) may be considered by the PSRT on a case-by-case basis, provided that the HgbA1c is ≤ 8% within the last 6 months (sites may draw these at screening).
4. Previous or current recipient of an investigational HIV vaccine (previous placebo/ control recipients are not excluded).
5. Receipt of non-HIV experimental vaccine(s) received within the last 1 year. Exceptions include vaccines that have subsequently undergone licensure or Emergency Use Authorization (EUA) by the FDA or World Health Organization (WHO) Emergency Use Listing (EUL), or if outside the US, by the national regulatory authority (RA) authorizing this clinical trial.
6. Congenital or acquired immunodeficiency, including systemic medication use likely to impair immune response to vaccine in the opinion of the site investigator, such as glucocorticoid use, equal to or greater than prednisone 10 mg/day within 3 months prior to enrollment.
7. Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
8. History of myocarditis and/or pericarditis.
9. Receipt of any vaccine within 4 weeks prior to enrollment.
10. Initiation of Ag-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval.
11. Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life of greater than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
12. History of serious reaction (eg, hypersensitivity, anaphylaxis) to any related vaccine or component of the study-vaccine regimen. Of note, the study proposed vaccine regimen includes components similar to components of the licensed COMIRNATY (Pfizer) and SPIKEVAX (Moderna) mRNA vaccines; severe reaction to these vaccines is therefore exclusionary.
13. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
14. Idiopathic urticaria within the past year.
15. Bleeding disorder diagnosed by a clinician which would make study procedures a contraindication.
16. Seizure disorder; febrile seizures as a child or seizures secondary to alcohol withdrawal more than 5 years ago are not exclusionary.
17. Asplenia or functional asplenia.
18. Active duty and reserve US military personnel.
19. Any other chronic or clinically significant condition that, in the clinical judgment of the investigator, would jeopardize the safety or rights of the study participant, including but not limited to: clinically significant forms of substance use or alcohol use disorder(s), serious psychiatric disorders, persons with any suicide attempt within the past 1 year (if between 1 and 2 years, consult PSRT for approval), or cancer that, in the clinical judgement of the site investigator, has potential for recurrence (excluding basal cell carcinoma).
20. Asthma is excluded if the participant has ANY of the following:

    * Required either oral or parenteral corticosteroids for an exacerbation 2 or more times within the past year; OR
    * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or coexisting conditions unrelated to asthma); OR
    * Uses a short-acting rescue inhaler more than 2 days/week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
    * Uses medium- to high-dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]); OR
    * Uses more than 1 medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than 1 medication for maintenance therapy daily for greater than 2 years requires PSRT approval.
21. A participant with a history of a potential immune-mediated medical condition (PIMMC), either active or remote. Not exclusionary: 1) Remote history of Bell's palsy (> 2 years ago) not associated with other neurologic symptoms and 2) Mild psoriasis or other mild, uncomplicated, localized or dermatologic condition that does not require ongoing systemic treatment.
22. History of allergy to local anesthetic (Novocaine, Lidocaine).
23. Investigator concern for difficulty with venous access based on clinical history and physical examination. For example, persons with a history of intravenous drug use or substantial difficulty with previous blood draws.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-07 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of local reactogenicity signs and symptoms after receipt of any study vaccine | Part A: Day 15, 71, and 127; Part B: Day 15, 71, 127, 183, and 239; Part C: 15, 71, 127, 183, and 239 (14 days following receipt of any study vaccine)
Frequency of systemic reactogenicity signs and symptoms after receipt of any study vaccine | Part A: Day 15, 71, and 127; Part B: Day 15, 71, 127, 183, and 239; Part C: 15, 71, 127, 183, and 239 (14 days following receipt of any study vaccine)
Number of serious adverse events (SAEs) leading to early participant withdrawal or permanent discontinuation | 31 months
Number of medically attended adverse events (MAAEs) leading to early participant withdrawal or permanent discontinuation | 31 months
Number of adverse events of special interest (AESIs) leading to early participant withdrawal or permanent discontinuation | 31 months
Number of adverse events (AEs) leading to early participant withdrawal or permanent discontinuation | 31 months
Part C only: Frequency of the CD4BS and CH505M5, G458Y, GNT1-specific, N280D KO IgG+ memory B cells, as assessed by flow cytometry | Part C: Day 127 and 239 (2 weeks after the third and fifth vaccinations respectively)
Part C only: Response rate of serum Ab neutralization of vaccine-matched tier 2 HIV-1 strains as measured by TZM-bl assay | Part C: Day 127 and 239 (2 weeks after the third and fifth vaccinations respectively)
Part C only: Magnitude of serum Ab neutralization of vaccine-matched tier 2 HIV-1 strains as measured by TZM-bl assay | Part C: Day 127 and 239 (2 weeks after the third and fifth vaccinations respectively)

SECONDARY OUTCOMES:
Parts B and C: Response rate of serum IgG binding Abs to autologous and heterologous HIV Env stabilized trimers, as assessed by binding antibody multiplex assay (BAMA) | Part B: Day 127 and 239; Part C: Day 127 and 239 (2 weeks after the third and fifth vaccinations, respectively, in each part)
Parts B and C: Magnitude of serum IgG binding Abs to autologous and heterologous HIV Env stabilized trimers, as assessed by binding antibody multiplex assay (BAMA) | Part B: Day 127 and 239; Part C: Day 127 and 239 (2 weeks after the third and fifth vaccinations, respectively, in each part)
Part B only: Response rate of serum Ab neutralization of vaccine-matched tier 2 HIV-1 strains as measured by the TZM-bl assay | Part B: Day 127 and 239 (2 weeks after the third and fifth vaccinations respectively)
Part B only: Magnitude of serum Ab neutralization of vaccine-matched tier 2 HIV-1 strains as measured by the TZM-bl assay | Part B: Day 127 and 239 (2 weeks after the third and fifth vaccinations respectively)
Parts B and C: Response rate of differential serum Ab neutralization of precursor detection virus and corresponding epitope KO virus, as measured by TZM-bl assay | Part B: Day 127 and 239; Part C: Day 127 and 239 (2 weeks after the third and fifth vaccinations, respectively, in each part)
Parts B and C: Magnitude of differential serum Ab neutralization of precursor detection virus and corresponding epitope KO virus, as measured by TZM-bl assay | Part B: Day 127 and 239; Part C: Day 127 and 239 (2 weeks after the third and fifth vaccinations, respectively, in each part)
Parts B and C: Response rate of serum Ab neutralization of heterologous HIV-1 strains, as measured by TZM-bl assay | Part B: Day 127 and 239; Part C: Day 127 and 239 (2 weeks after the third and fifth vaccinations, respectively, in each part)
Parts B and C: Magnitude of serum Ab neutralization of heterologous HIV-1 strains, as measured by TZM-bl assay | Part B: Day 127 and 239; Part C: Day 127 and 239 (2 weeks after the third and fifth vaccinations, respectively, in each part)
Parts B and C: Response rate of CD4+ and CD8+ T-cell responses, as measured by flow cytometry | Part B: Day 127 and 239; Part C: Day 127 and 239 (2 weeks after the third and fifth vaccinations, respectively, in each part)
Parts B and C: Magnitude of CD4+ and CD8+ T-cell responses, as measured by flow cytometry | Part B: Day 127 and 239; Part C: Day 127 and 239 (2 weeks after the third and fifth vaccinations, respectively, in each part)
Part B only: Frequency of the CD4BS and CH505M5, G458Y, GNT1-specific, N280D KO IgG+ memory B cells, as assessed by flow cytometry | Part B: Day 127 and 239 (2 weeks after the third and fifth vaccinations respectively)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Alabama CRS (Site ID: 31788), Birmingham, Alabama
  - The Ponce de Leon Center CRS (Site ID: 5802), Atlanta, Georgia
  - Vanderbilt Vaccine (VV) CRS (Site ID: 30352), Nashville, Tennessee
- South Africa (3):
  - Setshaba Research Centre CRS (Site ID: 31829), Soshanguve, Gauteng
  - Isipingo CRS (Site ID: 31635), Isipingo, KwaZulu-Natal
  - Klerksdorp CRS (Site ID: 30325), Klerksdorp, North West

IPD SHARING:
Plan to Share IPD: No